CLINICAL TRIAL: NCT06297161
Title: Post Marketing Surveillance Study to Observe Safety and Effectiveness of BOSULIF
Brief Title: A Study to Learn About the Study Medicine Bosulif in Adult Patients With Chronic Myeloid Leukemia(CML).
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1871065; NCT06297161 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Leukemia Myelogenous
Keywords: Philadelphia chromosome-positive (Ph+)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with newly diagnosed CP Ph+ CML: Patients newly-diagnosed with chronic phase (CP) Philadelphia chromosome-positive chronic myelogenous leukemia (Ph+ CML)
  Interventions: Drug: Bosulif

INTERVENTIONS:
Drug: Bosulif — chronic myelogenous leukemia patients

SUMMARY:
The purpose of this study is to look at how safe and effective is bosulif in routine clinical practice.

This study is seeking for participants who are:

* Adult Patients who are just confirmed to have Chronic Myeloid Leukemia (CML) defined in Local Product Document (LPD). CML is a type of cancer that starts in the blood-forming cells of the bone marrow and invades the blood. LPD explains what a medicine's benefits and problems are. LPD also explains how to use the medicine correctly in Korea.
* willing to take part in the study after being informed about the study. All participants in this study will receive bosulif. All participants who have entered this study should meet the usual prescribing criteria for bosulif as per the LPD. The participants will be treated with bosulif under routine clinical practice in Korea.

The study will look at the experiences of people receiving the study medicine. This will help to see if the study medicine is safe and effective.

In this study all treatment and checking of the patients will be done as per the study doctor. The study can be performed in Korean health care centers where bosulif is prescribed to treat CML after the patients have agreed to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients newly-diagnosed chronic phase (CP) Philadelphia chromosome-positive chronic myelogenous leukemia (Ph+ CML) or CP, AP, BP Ph+ CML with resistance or intolerance to prior therapy
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

- Patients to whom bosulif is contraindicated as per the local labeling- Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Newly-diagnosed chronic phase (CP) Philadelphia chromosome-positive chronic myelogenous leukemia (Ph+ CML) or Chronic phase, accelerated phase (AP), or blast phase (BP) Ph+ CML with resistance or intolerance to prior therapy who are administrated Bosulif according to the approval label in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | From the date of bosulif treatment completion until index period (Between 30 Dec 2022 and 29 Dec 2028)

SECONDARY OUTCOMES:
Hematologic response: CHR, not achieved | From the date of bosulif treatment completion until index period (Between 30 Dec 2022 and 29 Dec 2028)
Cytogenetic response: CCyR, PCyR, mCyR, not achieved | From the date of bosulif treatment completion until index period (Between 30 Dec 2022 and 29 Dec 2028)
Molecular response: EMR, MMR, MR4.0, MR4.5, not achieved | From the date of bosulif treatment completion until index period (Between 30 Dec 2022 and 29 Dec 2028)
Relapse after Bosulif response | From the date of bosulif treatment completion until index period (Between 30 Dec 2022 and 29 Dec 2028)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871065